CLINICAL TRIAL: NCT04033575
Title: Clinical Investigation of a Toothpaste Containing Stannous Fluoride as Compared to Colgate Fluoride Toothpaste in Reducing Plaque and Gingivitis - a Three Month Study
Brief Title: Clinical Investigation of a Toothpaste Containing Stannous Fluoride as Compared to Colgate Fluoride Toothpaste
Acronym: CP_Total
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2019-03-PG-SNF-FL-BGS
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Tin Fluorides; Centers for Disease Control and Prevention, U.S.

STUDY DESIGN:
Intervention Model Description: This was a 6-month, randomized, single-center, parallel group, double-blinded, clinical research study to assess the clinical efficacy of two toothpastes containing stannous fluoride (SnHW and CPH) as compared to Regular Fluoride Toothpaste on the reduction of established dental plaque and gingivitis in adults.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: CRO-2019-03-PG-SNF-FL-BGS Product XXX Brush your teeth twice daily (morning and evening) for two (2) minutes each time.
  Cover the length of the toothbrush bristles with the toothpaste. For investigational use only by the study participant. Not for sale. For Adult Use Only. Keep out of reach of children under 6 years.
  In case of emergency or for further information contact:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoride Control (Sham Comparator): Colgate Cavity Protection 0.76% as Na MFP Toothpaste
  Interventions: Drug: Colgate Cavity Protection toothpaste
- Colgate Total SF (Active Comparator): Colgate Total Clean Mint White Paste 1100 ppm F Toothpaste
  Interventions: Drug: Colgate Total SF

INTERVENTIONS:
Drug: Colgate Total SF — 1100 ppm F Colgate Total Clean Mint White Paste Toothpaste is a test treatment
  Other Names: Stannous Fluoride
  Arms: Colgate Total SF
Drug: Colgate Cavity Protection toothpaste — 0.76% monofluorophosphate (1000 ppm MFP), Colgate Cavity Protection toothpaste is a control treatment.
  Other Names: CDC
  Arms: Fluoride Control

SUMMARY:
The objective of this study is to evaluate the clinical efficacy of a toothpaste containing stannous fluoride as compared to Colgate Fluoride Toothpaste in reducing plaque and gingivitis - a three- month study.

DETAILED DESCRIPTION:
This was a 6-month, randomized, single-center, parallel group, double-blinded, clinical research study to assess the clinical efficacy of two toothpastes containing stannous fluoride (SnHW and CPH) as compared to Regular Fluoride Toothpaste on the reduction of established dental plaque and gingivitis in adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, ages 18-70, inclusive.
* Availability for the six-month duration ofthe clinical research study.
* Good general health.
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein °Plaque Index (Turesky Modification).
* Signed Informed Consent Form.

Exclusion Criteria:

* Presence of partial denture.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one month prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition which prohibits eating or drinking for periods up to 4 hours.
* History of alcohol or drug abuse.
* Pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Gingivitis Scores | Baseline
  Gingivitis scale (Loe & Silness Gingival Index) Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Gingivitis Scores | 3 months
  Gingivitis scale (Loe & Silness Gingival Index) Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Dental Plaque Score | Baseline
  Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Dental Plaque Score | 3 months
  Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)

CONTACTS AND LOCATIONS:
Overall Officials: Yun Po Zhang, Doctoral, Study Director — Colgate Palmolive
Locations (1):
- Consumer Research Consulting, LLC, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No